CLINICAL TRIAL: NCT00528099
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IMA-026 Administered Subcutaneously or Intravenously to Healthy Japanese Male Subjects
Brief Title: Study Evaluating IMA-026 in Healthy Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3192K1-1001
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: IMA-026 — SC and IV ascending single doses from lyophilized dosage form 0.3, 1, 2, 4 mg/kg SC and 3 mg/kg IV

SUMMARY:
To assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of ascending, single subcutaneous or intravenous doses of IMA-026 in healthy Japanese male subjects

ELIGIBILITY:
Inclusion Criteria:

* Men ages 20 to 40 years, inclusive, at screening
* Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight > 45 kg
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vitals signs, and 12 lead ECG.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and PK profile of IMA-026 administered as single ascending subcutaneous or intravenous doses. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Toshima-ku, Tokyo, Japan